CLINICAL TRIAL: NCT05529888
Title: Serum Homocysteine Level in Acne Patients Before and After Oral Isotretinoin
Brief Title: Measure the Serum Level of Homocysteine in Acne Patients Before and After Oral Isotretinoin.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Doaa Hamdi Abd Elal Mohamed, Principal Investigator, Aswan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 322/1/19
Record Dates: First submitted 2022-09-01; First posted 2022-09-07 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Isotretinoin

STUDY DESIGN:
Intervention Model Description: group of patients and group of control
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient group (Active Comparator): Patients were treated with Isotretinoin in a dose (from 20 to 40) for 3 months and serum homocysteine were assessed before and after treatment
  Interventions: Drug: Isotretinoin
- Control group (No Intervention): Assessment of serum YKL40 in healthy individuals

INTERVENTIONS:
Drug: Isotretinoin — Isotretinoin is a vitamin-A derivative for treatment of moderate to severe acne used in a dose from 20-40 mg for 3 months duration
  Arms: Patient group

SUMMARY:
Serum homocysteine level in Acne patients before and after oral Isotretinoin and Correlation between serum level of homocysteine in acne patients before and after Oral isotretinoin treatment

DETAILED DESCRIPTION:
Acne vulgaris is a common chronic inflammatory disease of the skin. It is found in about 80% of young adults and adolescents. It is a disease that affects the pilosebaceous units of the skin and may result in inflammatory or non-inflammatory lesions,Oral isotretinoin (13-cis-retinoic acid) is the only drug that counteracts all the pathogenetic mechanisms that contribute to the development of acne The standard dose of isotretinoin is 0.5 to 1 mg/kg per day for 4 months to a cumulative dose of 120-140 mg/kg is effective in the management of acne vulgaris The scope of our study is to detect serum homocysteine level in acne patient befor and after oral isotrtinoin treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes with acne vulgaris

Exclusion Criteria:

* Patients with history of malignancies.
* Patients with renal and hepatic dysfunction.
* Cardiac patient.
* Pregnant, lactating and female welling to have pregnancy in the period of study.
* Patient with absorption disorder.
* Patient with history of favism.
* Patient has already been treated with isotretinoin.

Ages: 15 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of oral isotretinoin on Serum homocysteine in acne vulgaris patients | 3 months
  Assessment in serum level homocysteine level in acne vulgaris patients after isotretinoin therapy with assesment of its level before starting therapy for detecting changes in serum homocysteine and effect of isotretinoin therapy on it.

CONTACTS AND LOCATIONS:
Locations (1):
- Aswan University-Faculty of Medicine, Aswān, New Aswan City, Egypt

IPD SHARING:
Plan to Share IPD: No